CLINICAL TRIAL: NCT05713786
Title: Effects of Physical Exercise and Motor Activity on Post-mastectomy Pain.
Brief Title: Physical Exercise, Motor Activity and Post-mastectomy Pain Syndrome.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Other Study IDs: BRCAMA
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Post mastectomy pain syndrome; Motor activity; Pain markers
MeSH Terms: conditions — Chronic Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Pain is an unpleasant sensation common to all those who undergo surgery. Several studies indicate that 40-60% of patients experience the post-operative experience and can be caused by both internal and external stimuli. The most patients define the post-operative experience as a very painful condition that interferes with normal daily activities. Chronic post mastectomy pain is a condition characterized by pain in the anterior chest, armpit, and/or upper arm, usually ipsilateral to surgery, which begins after mastectomy or quadrantectomy and persists for longer. three months after surgery. It can become chronic in a broad spectrum of conditions. In fact, it is estimated that between 10 and 50% of elective interventions can generate persistent post-surgical pain.

Aim of this prospective observational study is to evaluate the effects of motor and/or sports activity on the intensity and interference of chronic pain in quality of life of women underwent mastectomy.

DETAILED DESCRIPTION:
Acute post surgery pain is defined as a normal physiological response to an injurious stimulus.

Adequate monitoring associated with appropriate postoperative pain therapy significantly contribute to the improvement of perioperative morbidity, assessed in terms of lower incidence of postoperative complications. In addition, many patients undergo important changes in emotional and affective behavior: acute pain anxiety is often replaced by reactive depression and hypochondria combined with somatization and worsening of quality of life. The latter is an important factor in the context of tumor pathology. Since, while the goal of achieving 100% survival in women with breast cancer is still pursued, so too is improving the quality of life and restoring optimal levels of function of patients.The benefits of physical activity on the general population have been extensively studied. It has been shown that physical activity in the cancer patient allows the recovery of the previous functional capacities, strength and flexibility, improvement of the pain symptom and asthenia, as well as the reduction of alterations in the haematological picture such as neutropenia, anemia, thrombocytopenia.

Breast cancer is due to the uncontrolled multiplication of certain cells in the mammary gland which turn into malignant cells. The most frequent tumors arise from glandular cells (lobules) or from those that form the wall of the ducts.

Breast cancers can be invasive or non-invasive. The most invasive forms are usually ductal carcinoma, which affects the milk ducts beyond the duct wall and accounts for 70-80 percent of all forms of breast cancer, and lobular carcinoma that exceeds the wall of the lobule. Breast cancer is classified into 5 stages (0 to IV).

Chronic post mastectomy pain is a condition characterized by pain in the front of the chest, armpit, and / or upper arm, usually ipsilateral to surgery, which begins after mastectomy or quadrantectomy and persists for longer. three months after surgery (International Association for the Study of Pain.

In cancer patients, the level of pain intensity can be used in pain management as a subjective indicator to be quantitatively assessed together with what is defined as "interference of pain in activities of daily living". Interference is a key biomarker for establishing adequate pain therapy. Pain intensity and interference are both measured using questionnaires / scales such as the Numerical Rating Scale (NRS), the Brief Pain Inventory (BPI).

Finally, inflammatory responses and oxidative balance play key roles in the development and persistence of many pathological pain states. In light of the above, a prospective observational clinical study is proposed in order to evaluate the influence of motor activity on the intensity and interference of chronic pain in women who have undergone mastectomy surgery due to resection of stage breast cancer. II and III.

Study population: women underwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer not followed by breast reconstruction aged 18 years or older who have not received chemotherapy or radiation.

Pain assessment Pain assessment is a multidimensional process, which must take into account all the components of suffering, both physically, psychologically and socially. The assessment of pain and motor activity of each participant in the study will be carried out 3 and 6 months after surgery. Pain will be assessed by administration of the following questionnaires: Numerical Rating Scale, Brief Inventory Pain.

The IPAQ (International Physical Activity Questionnaire) questionnaire measures the type and amount of physical activity that is normally done. The questions refer to the activity carried out in the last 7 days. It will be administered at 3 and 6 months after surgery.The expected duration of the study can be considered to be approximately 12 months.

Interference is a key biomarker for establishing adequate pain therapy. Pain intensity and interference will be both measured using questionnaires/scales such as the numerical Rating scale (NRS), the Brief Pain Inventory (BPI) will be assessed 12 and 24 weeks after mastectomy by administration of the following questionnaires: Numerical Rating Scale, Brief Inventory Pain. Physical activity will be assessed by means of the IPAQ questionnaire (International Physical Activity.

At the same timepoints (12 and 24 weeks after surgery) biomarkers of pain, inflammation (C-reactive protein, Interleukin-6, interleukin-8, tumor necrosis factor-alpha) and oxidative stress (superoxide dismutase, catalase and malondyaldheide) will be measured together with routinary blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 with a diagnosis of previous Stages I-III breast cancer.

Exclusion Criteria:

* medical history of other types of cancer;
* disease related to the immune system (e.g. multiple sclerosis, HIV, lupus);
* recent symptoms of illness (cough, fever);
* waiting breast reconstruction;
* not chemotherapy or radiation during the first six months after surgery:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women underwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Effects of motor and/or sports activity on the intensity of chronic pain in women underwent mastectomy. | Evaluation performed three and six months after surgery
  Pain intensity self-measured using the Numerical Rating Scale (NRS). NRS is a 0-11 point-scale where the end points are the extremes of no pain (point 0) and worst pain as bad as it could be (point 10).
Effects of motor and/or sports activity on interference of chronic pain in women underwent mastectomy. | Evaluation performed three and six months after surgery
  Interference of pain in activities of daily living is a key biomarker for establishing adequate pain therapy. Interference of pain measured with the Brief Pain Inventory - Short Form. It is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily activities. Each item is scored on a 10 point numeric rating scale where 0 = no interference/pain and 10 = severe or complete interference/pain.

SECONDARY OUTCOMES:
Biomarkers of inflammation. | Evaluation performed three and six months after surgery
  Biomarkers of inflammation were evaluated in serum. Analysis was performed in blood aliquot withdrawn during the routinary exames. The following biomarkers were considered: C reactive protein (CRP), was evaluated by cytofluorimetry; intrleukin 6 (IL6), interleukin 8 (IL8), tumor necrosis factor alpha (TNFa) were evaluated by ELISA.
Biomarkers of oxidative stress | Evaluation performed three and six months after surgery
  Biomarkers of oxidative stress were evaluated in serum. Analysis was performed in blood aliquot withdrawn during the routinary exames. The following biomarkers of oxidative stress were considered: superoxide dismutase (SOD), catalase (CAT) and manlondialdheyde (MDA). SOD and CAT activity was evaluated by colorimetric assay, MDA by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Gioacchino Calapai, MD, Study Director — Azienda Ospedaliera Universitaria "G. Martino"
Locations (1):
- Gioacchino Calapai, Messina, Italy

REFERENCES:
- [Background] Calapai M, Esposito E, Puzzo L, Vecchio DA, Blandino R, Bova G, Quattrone D, Mannucci C, Ammendolia I, Mondello C, Gangemi S, Calapai G, Cardia L. Post-Mastectomy Pain: An Updated Overview on Risk Factors, Predictors, and Markers. Life (Basel). 2021 Sep 29;11(10):1026. doi: 10.3390/life11101026. PMID 34685397
- [Background] Ambrose KR, Golightly YM. Physical exercise as non-pharmacological treatment of chronic pain: Why and when. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):120-30. doi: 10.1016/j.berh.2015.04.022. Epub 2015 May 23. PMID 26267006
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Tait RC, Zoberi K, Ferguson M, Levenhagen K, Luebbert RA, Rowland K, Salsich GB, Herndon C. Persistent Post-Mastectomy Pain: Risk Factors and Current Approaches to Treatment. J Pain. 2018 Dec;19(12):1367-1383. doi: 10.1016/j.jpain.2018.06.002. Epub 2018 Jun 30. PMID 29966772
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Schug SA, Bruce J. Risk stratification for the development of chronic postsurgical pain. Pain Rep. 2017 Oct 31;2(6):e627. doi: 10.1097/PR9.0000000000000627. eCollection 2017 Nov. PMID 29392241
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Kaushik AS, Strath LJ, Sorge RE. Dietary Interventions for Treatment of Chronic Pain: Oxidative Stress and Inflammation. Pain Ther. 2020 Dec;9(2):487-498. doi: 10.1007/s40122-020-00200-5. Epub 2020 Oct 21. PMID 33085012